CLINICAL TRIAL: NCT01659736
Title: Transcranial Magnetic Stimulation Treatment for Generalized Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Neuronetics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIEF003523.1
Record Dates: First submitted 2012-05-25; First posted 2012-08-08 (Estimated); Results first posted 2016-01-07 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Generalized Anxiety Disorder
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TMS Therapy (Experimental): TMS treatment
  Interventions: Device: TMS
- TMS-Sham (Sham Comparator): This is a sham TMS condition
  Interventions: Device: TMS

INTERVENTIONS:
Device: TMS — Treatment will entail daily (5 days/week) sessions of TMS for 6 weeks.
  Other Names: Transcranial Magnetic Stimulation

SUMMARY:
This study is investigating a new indication of Transcranial Magnetic Stimulation (TMS) by conducting a pilot randomized-controlled trial (RCT) comparing structural neuronavigation-directed TMS to Sham-TMS Placebo therapy for treatment of Generalized Anxiety Disorder (GAD).

DETAILED DESCRIPTION:
Participants will complete structural MRI for neuronavigation. Participants will be randomly assigned to treatment condition. TMS or Sham-TMS sessions will occur daily 5 days/week for 6 weeks. Assessments will occur at pretreatment, weekly during treatment, post-treatment, and 3 month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with GAD as the principal or co-principal disorder
* Clinical Global Impression Score ≥ 4
* Hamilton Anxiety Rating Scale ≥ 18
* Hamilton Rating Scale for Depression ≤ 17
* Fluency in English
* Capacity to understand the nature of the study and willingness to sign informed consent form.

Exclusion Criteria:

* History of epilepsy or head trauma (LOC > 5 minutes) within the past 6 months.
* Lifetime history of increased intracranial pressure, seizure disorder, stroke, brain tumor, multiple sclerosis, or brain surgery.
* A review of patient medications by the study physician indicates an increased risk of seizure.
* An active autoimmune, endocrine, viral, or vascular disorder affecting the brain; any unstable cardiac disease; hypertension; or severe renal or liver insufficiency.
* Substance use disorder or PTSD within the past 6 months.
* Lifetime bipolar disorder, obsessive-compulsive disorder (OCD), psychotic disorder, mental retardation, or pervasive developmental disorder.
* Any psychotic features, including dementia or delirium. Concurrent psychotherapy and unwillingness to discontinue
* Medication change within past 3 months.
* Current serious suicidal or homicidal ideation, and/or serious suicidal attempt within past 6 months.
* Serious, unstable, or terminal medical condition or clinically judged too psychiatrically unstable to participate in the study.
* Any contraindication for participation in MRI scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen J Diefenbach, Ph.D., Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diefenbach GJ, Bragdon LB, Zertuche L, Hyatt CJ, Hallion LS, Tolin DF, Goethe JW, Assaf M. Repetitive transcranial magnetic stimulation for generalised anxiety disorder: a pilot randomised, double-blind, sham-controlled trial. Br J Psychiatry. 2016 Sep;209(3):222-8. doi: 10.1192/bjp.bp.115.168203. Epub 2016 May 19. PMID 27198484

RESULTS

PARTICIPANT FLOW:
Groups:
- TMS-Treatment: TMS treatment
  TMS: Treatment will entail daily (5 days/week) sessions of TMS for 6 weeks.
  Treatment in the substudy will entail 2 days/week sessions of TMS for 5 weeks.
- TMS-Sham: This is a sham TMS condition
  TMS: Treatment will entail daily (5 days/week) sessions of TMS for 6 weeks.
  Treatment in the substudy will entail 2 days/week sessions of TMS for 5 weeks.
Period: Treatment Period
Arm/Group | TMS-Treatment | TMS-Sham
Started | 14 | 12
Completed | 9 (n = 10, but data from one completer was excluded from all analyses due to protocol violation.) | 10
Not Completed | 5 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: 3-month Follow-up
Arm/Group | TMS-Treatment | TMS-Sham
Started | 9 | 10
Completed | 9 | 9
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- TMS Therapy: TMS treatment
  TMS: Treatment will entail daily (5 days/week) sessions of TMS for 6 weeks.
  Treatment in the substudy will entail 2 days/week sessions of TMS for 5 weeks.
- Total: Total of all reporting groups
Arm/Group | TMS Therapy | TMS-Sham | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.00 (11.95) | 44.58 (14.75) | 44.28 (13.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 13 | 12 | 25

OUTCOME MEASURES:

1. Primary Outcome: Change in the Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A) at Post-treatment and 3-month Follow-up.
Description: Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A) scores range from 0-56 with higher scores indicating more severe anxiety.
Time Frame: Pretreatment, Post-treatment (6 weeks after pretreatment), 3-month follow-up
Population: Intent-to-treat sample (n = 25)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | TMS-Treatment | TMS-Sham
Number analyzed (Participants) | 13 | 12
units on a scale
  pre-treatment | 25.31 (5.23) | 20.75 (3.72)
  post-treatment | 12.10 (5.77) | 14.38 (4.78)
  3-month follow-up | 10.36 (7.86) | 17.95 (7.48)
Statistical Analysis 1: Comparison: TMS-Treatment vs TMS-Sham; Test type: Superiority or Other; p = 0.006, ANOVA — p-value is for the condition (active TMS versus Sham) by time (pre, post, 3-month follow-up) interaction

2. Primary Outcome: Responder Status
Description: Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A) scores range from 0-56 with higher scores indicating more severe anxiety. Responder status was defined as a ≥ 50% improvement (i.e., reduction) in SIGH-A scores from pre-treatment to post-treatment.
Time Frame: Post-treatment, 6 weeks
Population: Post-treatment completers
Measure: Number; unit: participants
Groups:
- TMS- Treatment: TMS treatment
  TMS: Treatment will entail daily (5 days/week) sessions of TMS for 6 weeks.
  Treatment in the substudy will entail 2 days/week sessions of TMS for 5 weeks.
- TMS- Sham: This is a sham TMS condition
  TMS: Treatment will entail daily (5 days/week) sessions of TMS for 6 weeks.
  Treatment in the substudy will entail 2 days/week sessions of TMS for 5 weeks.
Arm/Group | TMS- Treatment | TMS- Sham
Number analyzed (Participants) | 9 | 10
participants | 7 | 2

3. Primary Outcome: Remission Status
Description: Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A) scores range from 0-56 with higher scores indicating more severe anxiety. Remission status was defined as a SIGH-A score < 8 and Clinical Global Impression Improvement score = 1 ("very much improved") or 2 ("much improved") at post-treatment.
Time Frame: post-treatment, 6 weeks
Population: Post-treatment completers
Measure: Number; unit: participants
Arm/Group | TMS-Treatment | TMS-Sham
Number analyzed (Participants) | 9 | 10
participants | 3 | 1

4. Primary Outcome: Responder Status
Description: Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A) scores range from 0-56 with higher scores indicating more severe anxiety. Responder status was defined as a ≥ 50% improvement (i.e., reduction) in SIGH-A scores from pre-treatment to 3-month follow-up.
Time Frame: 3-month follow-up
Population: 3-month follow-up completers
Measure: Number; unit: participants
Arm/Group | TMS-Treatment | TMS-Sham
Number analyzed (Participants) | 9 | 9
participants | 7 | 0

5. Primary Outcome: Remission Status
Description: Structured Interview Guide for the Hamilton Anxiety Rating Scale (SIGH-A) scores range from 0-56 with higher scores indicating more severe anxiety. Remission status was defined as a SIGH-A score < 8 and Clinical Global Impression Improvement score = 1 ("very much improved") or 2 ("much improved") at 3-month follow-up.
Time Frame: 3-month follow-up
Population: 3-month follow-up completers
Measure: Number; unit: participants
Arm/Group | TMS-Treatment | TMS-Sham
Number analyzed (Participants) | 9 | 9
participants | 6 | 0

ADVERSE EVENTS:
Arm/Group | TMS-Treatment | TMS-Sham
Serious Adverse Events (participants affected / at risk) | 1/13 | 0/12
Other Adverse Events (participants affected / at risk) | 13/13 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMS-Treatment (N=13) | TMS-Sham (N=12)
Chest Pain (Cardiac disorders) | 1 (1) | 0 (0) — A patient in the active group was hospitalized for evaluation of chest pain; however, the event was determined to be unrelated to the study intervention.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TMS-Treatment (N=13) | TMS-Sham (N=12)
Pin Prick Sensation (Nervous system disorders) | 9 | 10
Pain at the stimulation site (Nervous system disorders) | 11 | 8
Facial pain (including eye pain) (Nervous system disorders) | 3 | 1
Headache (Nervous system disorders) | 6 | 3
Toothache (Nervous system disorders) | 3 | 0
Lightheaded or Dizziness (Nervous system disorders) | 0 | 2
Facial twitch (Nervous system disorders) | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No